CLINICAL TRIAL: NCT04634734
Title: Correlation Between Periodontitis and Hypertension Among a Sample of Adult Egyptian Patients: A Hospital-based Cross-Sectional Study
Brief Title: Correlation Between Periodontitis and Hypertension Among a Sample of Adult Egyptian Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Saleh Yousef Al-Hasan, Principle Investigator, Cairo University
Other Study IDs: Correlation b/w Perio. & HBP
Record Dates: First submitted 2020-09-15; First posted 2020-11-18 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-09

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a cross-sectional study investigating the correlation between periodontitis and both hypertension and body mass index among a sample of adult Egyptian dental patients attending diagnostic center at faculty of Dentistry, Cairo University.

DETAILED DESCRIPTION:
* Dental patients will be recruited in a consecutive manner from the outpatient Diagnostic center, Faculty of Dentistry, Cairo University.
* Before the interview, the aim of the study will be explained to the patient and the patient's acceptance to participate in the survey will be received.
* Full questionnaire will be filled, then full mouth periodontal examination and charting will be done for each patient.
* The questionnaire will be filled through a face-to-face personal interview with the patient using simple, short, easily comprehended questions (Goulart A.C., Armani F. et al. 2017, Machado V., Aguilera E. M. et al. 2020). The questionnaire will be translated by a certified translator into Arabic and validated. All the interviews will be done by the same investigator.
* Non-respondent patients or patients refusing to participate will be reported with the cause of their refusal.
* The questionnaire which will be applied in study will include sociodemographic and medical questionnaires. These covariates will include gender, age, marital status (single, married/union of fact, divorced or widowed), occupation (student, employed, unemployed or retired) and smoking habits (current status: never, former, current). Education will be categorized according to the 2011 International Standard Classification of Education (ISCED-2011) (UNESCO 2012): no education (ISCED 0 level), elementary (ISCED 1-2 levels), middle (ISCED 3-4 levels), higher (ISCED 5- 8 levels) (ISCED 2011). Blood pressure will be measured at the clinic by automated sphygmomanometer device. Finally, measurements of height and weight will be taken at the clinical exam and body mass index (BMI) will be calculated as kg/m2.
* Clinical examination will be held on a dental unit using the light of the unit and a mirror. Periodontal status will be evaluated by full mouth charting using UNC 15 periodontal probe, including assessment of plaque index (PI), bleeding on probing (BOP), Probing Depth (PD), Clinical Attachment Level (CAL), gingival recession depth (Rec) and radiographic X-Ray imaging.
* Periodontitis case is defined according to the latest available EFP/AAP consensus. It will be defined if interdental CAL is detectable at ≥ 2 non-adjacent teeth, or buccal or oral CAL ≥ 3 mm with PPD > 3 mm at ≥ 2 teeth. Periodontitis staging will be defined according to severity and extent. Concerning severity, interdental CAL at the site of the greatest loss of 1-2 mm, 3-4 and ≥5 was considered as mild (Stage 1), moderate (Stage 2), and severe (Stage 3 and Stage 4), respectively (Tonetti, Greenwell et al. 2018).

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age is between 18-70 years old.
* Patients consulting in the outpatient clinic.
* Patients not receiving periodontal treatment within the previous four months.
* Provide informed consent.

Exclusion Criteria:

* Individuals with chronic systemic diseases such as endocrine, metabolic and hematological conditions.
* Patients having problem in opening their mouth or undergoing inter-maxillary fixation where oral examination will not be possible.
* Pregnant women.
* Patients diagnosed with psychiatric problems or intoxicated with alcohol or drugs.
* Patients consuming caffeine, doing exercise and smoking in the 30 min prior to blood pressure measurement.
* Third molars, dental implants and retained roots.
* Patients with orthodontic appliances.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Periodontitis adult patients with hypertension attending to diagnostic center at faculty of Dentistry, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between periodontitis and hypertension | Through study completion, an average of 1 year
  * Clinical examination will be held on a dental unit using the light of the unit and a mirror. Periodontal status will be evaluated by full mouth charting using UNC 15 periodontal probe, including assessment of plaque index (PI), bleeding on probing (BoP), Probing Depth (PD), Clinical Attachment Level (CAL) and digital radiographic imaging.
  * Periodontitis case is defined according to the latest available EFP/AAP consensus.
  * Blood pressure measured by using an automated sphygmomanometer device. hypertension will be defined as values of systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg, or; the use of antihypertensive medication.
  * Then a questionnaire will be collected to estimate the prevalence of hypertension in periodontitis Egyptians adult patients.

SECONDARY OUTCOMES:
Body mass index. | Through study completion, an average of 1 year
  to estimate the impact of overweight and obesity in periodontitis cases by body mass index (BMI); which is calculated as the body weight (kg) divided by the square of the height (m).